CLINICAL TRIAL: NCT02372409
Title: A Pilot Study of Using MRI-Guided Laser Heat Ablation to Induce Disruption of the Peritumoral Blood Brain Barrier to Enhance Delivery and Efficacy of Treatment of Pediatric Brain Tumors
Brief Title: Using MRI-Guided Laser Heat Ablation to Induce Disruption of the Peritumoral Blood Brain Barrier to Enhance Delivery and Efficacy of Treatment of Pediatric Brain Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accruals and competing clinical trials
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201502062
Record Dates: First submitted 2015-02-13; First posted 2015-02-26 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Glioma; Pilocytic Astrocytoma; Anaplastic Astrocytoma; Glioblastoma; Mixed Oligoastrocytoma; Mixed Glioma; Oligodendroglioma; Optic Glioma; Astrocytoma
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma; Oligodendroglioma; Optic Nerve Glioma | interventions — Doxorubicin; Etoposide; etoposide phosphate; Dynamic Contrast Enhanced Magnetic Resonance Imaging; Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A (MRI-guided laser ablation) (Experimental): * MLA is a minimally invasive laser surgery currently FDA approved for cytoreductive treatment of brain tumors, both primary and metastatic. MLA employs a small incision in the scalp and skull, through which a thin laser probe is inserted and guided by MR imaging to the core of a tumor mass where it delivers hyperthermic ablation from the core to the rim.
  * Participants will undergo DCE and DSC-MRI imaging at the following time points:
    * no more than 3 weeks prior to MLA (OPTIONAL)
    * within approximately 4 days after MLA
    * 2-4 weeks after MLA
    * Every 12 weeks (+/- 7 days) for the first year or until disease progression
  Interventions: Device: MRI-guided laser ablation; Device: Dynamic contrast-enhanced (DCE) MRI; Device: Dynamic susceptibility contrast (DSC) MRI
- Arm B (MRI-guided laser ablation, doxorubicin, etoposide) (Experimental): * MLA is a minimally invasive laser surgery currently FDA approved for cytoreductive treatment of brain tumors, both primary and metastatic. MLA employs a small incision in the scalp and skull, through which a thin laser probe is inserted and guided by MR imaging to the core of a tumor mass where it delivers hyperthermic ablation from the core to the rim.
  * Within 7 days of MLA (range 2-14 days) doxorubicin will be given intravenously on an outpatient basis weekly for 6 weeks at a dose of 25 mg/m^2 over 5-30 minutes
  * Following the completion of doxorubin, etoposide 50 mg/m^2/day will be given orally for 21 days of each 28-day cycle (treatment can continue up to 24 cycles)
  * Participants will undergo DCE and DSC-MRI imaging at the following time points:
    * no more than 3 weeks prior to MLA (OPTIONAL)
    * within approximately 4 days after MLA
    * 2-4 weeks after MLA
    * every 8 weeks (+/- 7 days) until 2 years have elapsed or disease progression, whichever comes first
  Interventions: Device: MRI-guided laser ablation; Drug: Doxorubicin; Drug: Etoposide; Device: Dynamic contrast-enhanced (DCE) MRI; Device: Dynamic susceptibility contrast (DSC) MRI

INTERVENTIONS:
Device: MRI-guided laser ablation
  Other Names: MLA
Drug: Doxorubicin
  Other Names: Adriamycin
  Arms: Arm B (MRI-guided laser ablation, doxorubicin, etoposide)
Drug: Etoposide
  Other Names: Etoposide phosphate; VP-16; Toposar; Etopophos; VePesid
  Arms: Arm B (MRI-guided laser ablation, doxorubicin, etoposide)
Device: Dynamic contrast-enhanced (DCE) MRI
  Other Names: DCE-MRI
Device: Dynamic susceptibility contrast (DSC) MRI
  Other Names: DSC-MRI

SUMMARY:
By employing a combination of advanced MRI techniques and correlative serum biomarkers of blood brain barrier (BBB) disruption, the investigators plan to develop a powerful, first of its kind clinical algorithm in pediatrics whereby the investigators can measure and identify the window of maximal BBB disruption post MLA to 1) allow for an alternative to surgery in incompletely resected tumors, 2) allow for optimal chemotherapeutic dosing to achieve the greatest benefits and the least systemic side effects and 3) distinguish subsequent tumor progression from long-term MLA treatment effects. Preliminary data in adult imaging studies have shown that the BBB disruption lasts for several weeks following treatment before returning to a low baseline. This pilot therapeutic study will provide preliminary validation in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

ARM A

* Presumed pediatric gliomas (grades I-IV) on MRI that are determined to be candidates for MLA by the treating neurosurgeon
* Age 3 to ≤ 21
* Karnofsky/Lansky performance status ≥ 60%

ARM B

* Recurrent pediatric brain tumors determined candidates for MLA as determined by the treating neurosurgeon.
* Unequivocal evidence of tumor progression by MRI
* There must be an interval of at least 12 weeks from the completion of radiotherapy to study registration except if there is unequivocal evidence for tumor recurrence per RANO criteria. When the interval is less than 12 weeks from the completion of radiotherapy, the use of PET scan is allowed to differentiate between evidence of tumor recurrence and pseudoprogression.
* Recurrent lesions with dimension and contour that are determined by the treating neurosurgeon to be appropriate for MLA.
* Age 3 to ≤ 21
* Karnofsky/Lansky performance status ≥ 60%
* Adequate cardiac function as determined by a shortening fraction ≥ 27% or left ventricular ejection fraction ≥ 50% by echocardiogram within the past 1 year prior to registration.
* Prior anthracycline therapy does not exceed 200 mg/m^2 total cumulative dose.
* Adequate bone marrow and hepatic function as defined below (must be within 7 days of MLA):

  * Absolute neutrophil count (ANC) ≥ 1000/mcl (G-CSF is allowed)
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 9 g/dL (pRBC transfusion +/- ESA are allowed)
  * ALT ≤ 3 x ULN
  * AST ≤ 3 x ULN
  * ALP ≤ 3 x ULN. If ALP is > 3 x ULN, GGT must be checked and be ≤ 3 x ULN.
  * Bilirubin ≤ 2 x ULN
* At the time of registration, patient must have recovered from the toxic effects of prior therapy to no more than grade 1 toxicity.
* At the time of registration, patient must be at least 4 weeks from other prior cytotoxic chemotherapy.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

ARM A

* Currently receiving or scheduled to receive any other therapies intended to treat the newly diagnosed glioma prior to MLA and the first post-MLA blood collection for correlative studies.
* Multi-focal or metastatic disease.
* Pregnant and/or breastfeeding. Premenopausal women must have a negative serum or urine pregnancy test within 14 days of study entry.
* Inability to undergo MRI due to personal or medical reasons.
* Known history of HIV or autoimmune diseases requiring immunosuppressant drugs.

ARM B

* Prior treatment with bevacizumab within 12 weeks of study entry.
* Previous treatment with complete cumulative doses of daunorubicin, idarubicin, and/or other anthracyclines and anthracenediones that is equivalent to a total dose of > 200 mg/m2 doxorubicin.
* More than 2 prior relapses (not counting the current relapse being treated on this study).
* Currently receiving any other investigational agents that are intended as treatments of the relapsed tumor.
* Multi-focal or metastatic disease.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to doxorubicin or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, recent heart attack within the previous 12 months or severe heart problems, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Premenopausal women must have a negative serum or urine pregnancy test within 14 days of study entry.
* Inability to undergo MRI due to personal or medical reasons.
* Known history of HIV or autoimmune diseases requiring immunosuppressant drugs.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cluster, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holodny AI, Nusbaum AO, Festa S, Pronin IN, Lee HJ, Kalnin AJ. Correlation between the degree of contrast enhancement and the volume of peritumoral edema in meningiomas and malignant gliomas. Neuroradiology. 1999 Nov;41(11):820-5. doi: 10.1007/s002340050848. PMID 10602854
- [Background] Kassner A, Thornhill R. Measuring the integrity of the human blood-brain barrier using magnetic resonance imaging. Methods Mol Biol. 2011;686:229-45. doi: 10.1007/978-1-60761-938-3_10. PMID 21082374
- [Background] Hawasli AH, Ray WZ, Murphy RK, Dacey RG Jr, Leuthardt EC. Magnetic resonance imaging-guided focused laser interstitial thermal therapy for subinsular metastatic adenocarcinoma: technical case report. Neurosurgery. 2012 Jun;70(2 Suppl Operative):332-7; discussion 338. doi: 10.1227/NEU.0b013e318232fc90. PMID 21869722
- [Background] Gong W, Wang Z, Liu N, Lin W, Wang X, Xu D, Liu H, Zeng C, Xie X, Mei X, Lu W. Improving efficiency of adriamycin crossing blood brain barrier by combination of thermosensitive liposomes and hyperthermia. Biol Pharm Bull. 2011;34(7):1058-64. doi: 10.1248/bpb.34.1058. PMID 21720013
- [Background] Quick J, Gessler F, Dutzmann S, Hattingen E, Harter PN, Weise LM, Franz K, Seifert V, Senft C. Benefit of tumor resection for recurrent glioblastoma. J Neurooncol. 2014 Apr;117(2):365-72. doi: 10.1007/s11060-014-1397-2. Epub 2014 Feb 15. PMID 24535317
- [Background] Ashley DM, Meier L, Kerby T, Zalduondo FM, Friedman HS, Gajjar A, Kun L, Duffner PK, Smith S, Longee D. Response of recurrent medulloblastoma to low-dose oral etoposide. J Clin Oncol. 1996 Jun;14(6):1922-7. doi: 10.1200/JCO.1996.14.6.1922. PMID 8656261
- [Background] Davidson A, Gowing R, Lowis S, Newell D, Lewis I, Dicks-Mireaux C, Pinkerton CR. Phase II study of 21 day schedule oral etoposide in children. New Agents Group of the United Kingdom Children's Cancer Study Group (UKCCSG). Eur J Cancer. 1997 Oct;33(11):1816-22. doi: 10.1016/s0959-8049(97)00201-3. PMID 9470839
- [Background] Fulton D, Urtasun R, Forsyth P. Phase II study of prolonged oral therapy with etoposide (VP16) for patients with recurrent malignant glioma. J Neurooncol. 1996 Feb;27(2):149-55. doi: 10.1007/BF00177478. PMID 8699237
- [Background] Law M, Young R, Babb J, Rad M, Sasaki T, Zagzag D, Johnson G. Comparing perfusion metrics obtained from a single compartment versus pharmacokinetic modeling methods using dynamic susceptibility contrast-enhanced perfusion MR imaging with glioma grade. AJNR Am J Neuroradiol. 2006 Oct;27(9):1975-82. PMID 17032878
- [Background] Blyth BJ, Farhavar A, Gee C, Hawthorn B, He H, Nayak A, Stocklein V, Bazarian JJ. Validation of serum markers for blood-brain barrier disruption in traumatic brain injury. J Neurotrauma. 2009 Sep;26(9):1497-1507. doi: 10.1089/neu.2008.0738. PMID 19257803
- [Background] Dunn GP, Dunn IF, Curry WT. Focus on TILs: Prognostic significance of tumor infiltrating lymphocytes in human glioma. Cancer Immun. 2007 Aug 13;7:12. PMID 17691714
- [Background] Dunn GP, Fecci PE, Curry WT. Cancer immunoediting in malignant glioma. Neurosurgery. 2012 Aug;71(2):201-22; discussion 222-3. doi: 10.1227/NEU.0b013e31824f840d. PMID 22353795
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (MRI-guided Laser Ablation) | Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide)
Started | 5 | 1
Completed | 3 | 0
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Disease progression | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (MRI-guided Laser Ablation) | Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide) | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Continuous [Median (Full Range); unit: years] | 11 [4 to 15] | 12 [12 to 12] | 11.5 [4 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Arm A Only: Number of Participants With Progression-free Survival (PFS)
Description: PFS is followed from start of treatment to time of progression or death, whichever occurs first.
Time Frame: Up to 5 years from date of registration (median length of follow-up, full range 196 days-1801 days)
Population: This outcome measure is for Arm A participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (MRI-guided Laser Ablation) | Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide)
Number analyzed (Participants) | 5 | 0
Participants | 4 |

2. Primary Outcome: Arm A Only: Overall Survival (OS) as Measured by Number of Participants Alive at 5 Years
Time Frame: Up to 5 years from date of registration (median length of follow-up, full range 196 days-1801 days)
Population: This outcome measure is for Arm A participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (MRI-guided Laser Ablation) | Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide)
Number analyzed (Participants) | 5 | 0
Participants | 5 |

3. Primary Outcome: Arm B Only: Number of Participants With Progression-free Survival (PFS)
Description: PFS is followed from start of treatment to time of progression or death, whichever occurs first.
Time Frame: At 6 months
Population: This outcome measure is for Arm B participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (MRI-guided Laser Ablation) | Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide)
Number analyzed (Participants) | 0 | 1
Participants |  | 0

4. Secondary Outcome: Change in Quality of Life as Measured by Karnofsky or Lansky Performance Status
Description: Score ranges from 100% to 10%. A higher score indicates that the patient has a more normal quality of life.
Time Frame: At 1 year post-MLA
Population: This data was not collected on the patient from Arm B.
Measure: Number; unit: score on a scale
Groups:
- Patient 1: Arm A (MRI-guided Laser Ablation); Patient 2: Arm A (MRI-guided Laser Ablation); Patient 3: Arm A (MRI-guided Laser Ablation); Patient 4: Arm A (MRI-guided Laser Ablation); Patient 5: Arm A (MRI-guided Laser Ablation): * MLA is a minimally invasive laser surgery currently FDA approved for cytoreductive treatment of brain tumors, both primary and metastatic. MLA employs a small incision in the scalp and skull, through which a thin laser probe is inserted and guided by MR imaging to the core of a tumor mass where it delivers hyperthermic ablation from the core to the rim.
  * Participants will undergo DCE and DSC-MRI imaging at the following time points:
    * no more than 3 weeks prior to MLA (OPTIONAL)
    * within approximately 4 days after MLA
    * 2-4 weeks after MLA
    * Every 12 weeks (+/- 7 days) for the first year or until disease progression
Arm/Group | Patient 1: Arm A (MRI-guided Laser Ablation) | Patient 2: Arm A (MRI-guided Laser Ablation) | Patient 3: Arm A (MRI-guided Laser Ablation) | Patient 4: Arm A (MRI-guided Laser Ablation) | Patient 5: Arm A (MRI-guided Laser Ablation)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
score on a scale
  Baseline | 90 | 100 | 80 | 100 | 100
  1 year post-MLA | 90 | 100 | 80 | 100 | 100

5. Secondary Outcome: Serum Biomarkers of Peritumoral Blood Brain Barrier (BBB) Disruption as Measured by Change in Neuron-specific Enolase (NSE)
Description: * Arm A patients had blood drawn at the following time points: baseline, 3 days post-MLA, 2-4 weeks post-MLA, and every 12 weeks thereafter for 12 months post-MLA
  * Arm B patients had blood drawn at the following time points: baseline, 3 days post-MLA, week 1, week 2, week 3, week 4, week 5, week 6, and every 8 weeks for the first 2 years or until disease progression, whichever occurs first.
  * Neuron specific enolase is an enzyme involved in glycolysis, which is localized in neurons and axonal processes. Potentially, it escapes into the blood and CSF at the time of neural injury. Elevated serum NSE seemed to correlates with disruption in BBB following MLA and transient increase in BBB permeability.
Time Frame: Up to 48 weeks post MRI-guided laser heat ablation (Arm A) or up to 2 years post MRI-guided laser heat ablation (Arm B)
Population: The one participant in Arm B did not consent to any procedures past 12 months post-MLA. There are time points not included because either the NSE was not detected in the samples or the samples were not collected.
Measure: Number; unit: ng/ml
Groups:
- Patient 6: Arm A (MRI-guided Laser Ablation): * MLA is a minimally invasive laser surgery currently FDA approved for cytoreductive treatment of brain tumors, both primary and metastatic. MLA employs a small incision in the scalp and skull, through which a thin laser probe is inserted and guided by MR imaging to the core of a tumor mass where it delivers hyperthermic ablation from the core to the rim.
  * Participants will undergo DCE and DSC-MRI imaging at the following time points:
    * no more than 3 weeks prior to MLA (OPTIONAL)
    * within approximately 4 days after MLA
    * 2-4 weeks after MLA
    * Every 12 weeks (+/- 7 days) for the first year or until disease progression
- Patient 1: Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide): * MLA is a minimally invasive laser surgery currently FDA approved for cytoreductive treatment of brain tumors, both primary and metastatic. MLA employs a small incision in the scalp and skull, through which a thin laser probe is inserted and guided by MR imaging to the core of a tumor mass where it delivers hyperthermic ablation from the core to the rim.
  * Within 7 days of MLA (range 2-14 days) doxorubicin will be given intravenously on an outpatient basis weekly for 6 weeks at a dose of 25 mg/m^2 over 5-30 minutes
  * Following the completion of doxorubin, etoposide 50 mg/m^2/day will be given orally for 21 days of each 28-day cycle (treatment can continue up to 24 cycles)
  * Participants will undergo DCE and DSC-MRI imaging at the following time points:
    * no more than 3 weeks prior to MLA (OPTIONAL)
    * within approximately 4 days after MLA
    * 2-4 weeks after MLA
    * every 8 weeks (+/- 7 days) until 2 years have elapsed or disease progression, whichever comes first
Arm/Group | Patient 1: Arm A (MRI-guided Laser Ablation) | Patient 4: Arm A (MRI-guided Laser Ablation) | Patient 3: Arm A (MRI-guided Laser Ablation) | Patient 5: Arm A (MRI-guided Laser Ablation) | Patient 6: Arm A (MRI-guided Laser Ablation) | Patient 1: Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1
ng/ml
  Baseline | 29.0219 | 58.3406 | 3.1823 | 13.1819 | 7.5534 | 11.5114
  Day 3 | 47.2666 | 26.7537 | 6.0443 | 33.8034 | 17.4680 | 18.5711
  1 week: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  1 week |  |  |  |  |  | 11.5909
  2 week: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  2 week |  |  |  |  |  | 8.6069
  2-4 weeks: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 0
  2-4 weeks | 12.0186 | 53.2519 | 5.4452 | 11.4998 | 9.3916 |
  4 week: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  4 week |  |  |  |  |  | 5.7440
  12 weeks: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 0
  12 weeks | 105.7828 | 15.1011 | 7.5436 | 206.8570 | 13.5989 |
  14 weeks: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  14 weeks |  |  |  |  |  | 6.1692
  24 weeks: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 0
  24 weeks | 19.1706 | 7.8464 | 3.8632 | 5.5086 | 13.8210 |
  36 weeks: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 0
  36 weeks | 22.8186 | 7.9655 |  | 10.0722 | 5.9368 |
  48 weeks: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 0
  48 weeks | 15.4708 | 35.6507 |  | 25.8530 | 5.9343 |

6. Secondary Outcome: Serum Biomarkers of Peritumoral Blood Brain Barrier (BBB) Disruption as Measured by Change in S100B
Description: * Arm A patients had blood drawn at the following time points: baseline, 3 days post-MLA, 2-4 weeks post-MLA, and every 12 weeks thereafter for 12 months post-MLA
  * Arm B patients had blood drawn at the following time points: baseline, 3 days post-MLA, week 1, week 2, week 3, week 4, week 5, week 6, and every 8 weeks for the first 2 years or until disease progression, whichever occurs first.
  * S100b is a low-molecular-weight Calcium-binding protein primarily found in astrocytic glial cells of the CNS. It is secreted by astrocytes for neuroprotective and -trophic cellular functions in the CNS. Elevated serum values can be associated with temporal changes in BBB integrity following MLA.
Time Frame: Up to 48 weeks post MRI-guided laser heat ablation (Arm A) or up to 2 years post MRI-guided laser heat ablation (Arm B)
Population: The one participant in Arm B did not consent to any procedures past 12 months post-MLA. There are time points not included because either the S100B was not detected in the samples or the samples were not collected.
Measure: Number; unit: pg/ml
Arm/Group | Patient 1: Arm A (MRI-guided Laser Ablation) | Patient 4: Arm A (MRI-guided Laser Ablation) | Patient 3: Arm A (MRI-guided Laser Ablation) | Patient 5: Arm A (MRI-guided Laser Ablation) | Patient 6: Arm A (MRI-guided Laser Ablation) | Patient 1: Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide)
Number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 1
pg/ml
  Baseline: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Baseline |  | 79.74 |  |  |  |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 1
  Day 3 | 39.90 | 58.86 |  |  |  | 35.90
  2-4 weeks: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  2-4 weeks |  | 55.74 |  |  |  |
  12 weeks: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 0
  12 weeks | 156.00 | 59.78 |  | 239.13 |  |
  24 weeks: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  24 weeks |  | 65.91 |  |  |  |
  36 weeks: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  36 weeks |  | 55.66 |  |  |  |
  48 weeks: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  48 weeks |  | 79.11 |  |  |  |

7. Secondary Outcome: Serum Biomarkers of Peritumoral Blood Brain Barrier (BBB) Disruption as Measured by Change in GFAP
Description: * Arm A patients had blood drawn at the following time points: baseline, 3 days post-MLA, 2-4 weeks post-MLA, and every 12 weeks thereafter for 12 months post-MLA
  * Arm B patients had blood drawn at the following time points: baseline, 3 days post-MLA, week 1, week 2, week 3, week 4, week 5, week 6, and every 8 weeks for the first 2 years or until disease progression, whichever occurs first.
  * The glial fibrillary acidic protein (GFAP) is a classic intermediate filament protein specific to astrocytes in the CNS. GFAP is characteristic of astrocyte- and neural stem cell-derived gliomas in CNS tumors and is used to identify malignancies of glial origin, such as astrocytomas and GBM. Serum GFAP values can be increased with temporal disruption of BBB post-MLA.
Time Frame: Up to 48 weeks post MRI-guided laser heat ablation (Arm A) or up to 2 years post MRI-guided laser heat ablation (Arm B)
Population: The one participant in Arm B did not consent to any procedures past 12 months post-MLA. There are time points not included because either the GFAP was not detected in the samples or the samples were not collected.
Measure: Number; unit: ng/ml
Arm/Group | Patient 1: Arm A (MRI-guided Laser Ablation) | Patient 4: Arm A (MRI-guided Laser Ablation) | Patient 3: Arm A (MRI-guided Laser Ablation) | Patient 5: Arm A (MRI-guided Laser Ablation) | Patient 6: Arm A (MRI-guided Laser Ablation) | Patient 1: Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide)
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 1
ng/ml
  Baseline: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Day 3 | 4.7370968 |  | 1.6146649 | 0.2225989 |  | 5.6051762
  2-4 weeks: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  2-4 weeks | 0.0652591 |  |  |  |  |
  12 weeks: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  24 weeks: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  36 weeks: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  48 weeks: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Correlation of MR Imaging With Peritumoral BBB Disruption
Description: The linear regression model will used to investigate the correlation between MR imaging and peritumoral BBB disruption. To account for correlation among the repeated measures from the same patient, the longitudinal data will be analyzed with the use of linear generalized estimating equation (GEE). Whether the average measurements differ at the multiple time points will be evaluated through GEE model. Least-square means at each time points will be presented and standard errors will be calculated within the use of the GEE sandwich method when accounting for within-patient correlation.
Time Frame: 1 year from MLA
Population: Data was not collected for this outcome measure.
Arm/Group | Arm A (MRI-guided Laser Ablation) | Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Predictive Value of the Peritumoral Permeability Score for Patient Outcome as Measured by PFS
Description: Biomarkers with higher correlation coefficient (r approaching 1) will be given higher priority. A minimum r=0.5 is required for inclusion for further analysis and will be used as a peritumoral permeability score. This score will then be correlated with the patient outcome data (as measured by 6 month PFS rate) to determine whether it has a predictive value.
Time Frame: 6 months
Population: Data was not collected for this outcome measure.
Arm/Group | Arm A (MRI-guided Laser Ablation) | Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: -Reportable adverse events will be tracked for 30 days following the last day of study treatment for patients in Arm B and for 30 days following the MLA for patients in Arm A. -All-cause mortality will be collected from start of treatment up to 5 years after start of treatment (median length of follow-up 413.5 days, full range 366 days-1801 days).
Description: For patients in Arm A, adverse events (of any grade) considered possibly, probably, or definitely related to the MLA need be reported. Adverse events that are possibly, probably, or definitely related to study procedures will be followed until resolution or stabilization of the event. "Stabilization" is defined as remaining at a consistent CTCAE version 4.0 grade of the event for two consecutive assessments. For Arm B, all grade 3 and higher events regardless of attribution are to be reported.
Arm/Group | Arm A (MRI-guided Laser Ablation) | Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/1
Other Adverse Events (participants affected / at risk) | 5/5 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (MRI-guided Laser Ablation) (N=5) | Arm B (MRI-guided Laser Ablation, Doxorubicin, Etoposide) (N=1)
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Noise sensitive (Social circumstances) | 1 | 0

LIMITATIONS AND CAVEATS:
The protocol stated that participants were to be followed for 5 years from participant registration or until death, whichever occurred first. The original consent that the participants signed stated that they would only be followed for 12 months after MLA. Once this issue was discovered, participants were contacted to be reconsented to be followed for 5 years; however, not all participants were able to be reconsented and that is why the results are late.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT02372409/Prot_SAP_000.pdf